CLINICAL TRIAL: NCT04977440
Title: High Protein Intake During the Early Phase of Critical Illness Compared With Normal Protein Intake
Brief Title: High Protein Intake in Critically Ill Ventilated Patients
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Farouk, lecturer, Cairo University
Other Study IDs: MS 29-2020
Record Dates: First submitted 2021-07-13; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Intensive Care Unit Syndrome
MeSH Terms: interventions — Whey Proteins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- standard protein
- high protein
  Interventions: Dietary Supplement: Whey protein

INTERVENTIONS:
Dietary Supplement: Whey protein — Patients were randomly divided into two groups: Group (A): Enteral feeding with normal protein intake ( 1.0 gm pin /kg/day ) Group (B): Enteral feeding with high protein intake ( 1.5- gm open /kg/day ) -Patient's- nonprotein- caloric intake was calculated according to REE :(25xactual body weight in kg ) and received it as follow : 1/2 the calculated amount of caloric intake in DAY 1 3/4 of the calculated amount of caloric intake in DAY 2
  -Full calculated caloric amount in DAY 3
  This regimen was followed long as the patient was tolerating the amount of feeding, and in case of intolerance:
  The volume of feeding boluses was decreased or Increase the time interval between boluses or IV metoclopramide or erythromycin was given
  Groups: high protein

SUMMARY:
This prospective interventional randomized control study was conducted on forty patients with respiratory failure; all patients were intubated and mechanically ventilated for at least three days. Twenty patients received high protein intake using whey protein, with daily follow-up of the blood sugar level, serum electrolytes, and chemistry. ICU outcome regarding food intolerance, 30-day mortality, length of MV and ICU-stay was recorded

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Mechanically ventilated patients (for three days or more )

Exclusion Criteria:

* Age < 18 years old
* Contraindication for enteral nutrition (gut ischemia, obstruction, or perforation)
* Expected intolerance for enteral nutrition (paralytic ileus)
* Inability to start enteral nutrition within 24-hours(i.e. surgery or other interventions)
* Short bowel syndrome
* Hemodynamic instability ( i.e shock state, need for vasopressors )
* Child C liver cirrhosis or acute liver failure
* Dialysis dependency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult mechanically ventilated patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Effect of high protein intake on glycemic control | up to 7 days
  measurements of blood glucose levels regularly after high protein intake
Effect of high protein intake on serum electrolytes | up to 7 days
  measurements of Na, K, Mg, phosphorous and calcium levels regularly after high protein intake

SECONDARY OUTCOMES:
Effect of high protein intake on ICU outcome | up to 7 days
  ICU outcome includes ICU survival , mechanical ventilation , food intolerance

CONTACTS AND LOCATIONS:
Overall Officials: farouk faris, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided